CLINICAL TRIAL: NCT07089602
Title: A Multicenter, Prospective, Randomized Controlled Modified Multi- Platform Trial Assessing the Efficacy of Human Placental Membrane Products and Standard of Care Versus Standard of Care Alone in the Management of Nonhealing Diabetic Foot Ulcers and Venous Leg Ulcers
Brief Title: Trial Assessing the Efficacy of Human Placental Membrane Products and Standard of Care Versus Standard of Care Alone in the Management of Nonhealing Diabetic Foot Ulcers and Venous Leg Ulcers
Acronym: BIOCAMP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: BioLab Holdings (Industry)
Collaborators: SerenaGroup, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIOCAMP
Record Dates: First submitted 2025-06-30; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Foot; DFU; Diabetic Foot Ulcer; Foot Ulcer, Diabetic; Ulcer Foot; Venous Leg Ulcer; Leg Ulcer; Leg Ulcers Venous; Ulcer
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer; Varicose Ulcer; Leg Ulcer; Ulcer

STUDY DESIGN:
Intervention Model Description: This study is a multi-center, prospective, randomized controlled clinical study consisting of 650 subjects from up to 30 centers. The subjects are randomized to receive 1 of 4 treatments, either with Tri-Membrane Wrap™ (HPM-1); Membrane Wrap™ (HPM-2); Membrane Wrap-Lite™ (HPM-3); Membrane Wrap-Hydro™ (HPM-4); and SOC. The target ulcers are evaluated weekly by the investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- DFU Standard of Care (Active Comparator): Debridement, reduction of bacterial burden, and proper moisture balance using dressings. Off-loading using the off-loading boot or total contact cast (TCC).
  Interventions: Other: Standard of Care DFU
- DFU Tri-Membrane Wrap™ + SOC (Experimental): Membrane Wrap-Lite™ is an allograft derived from human amniotic membrane.
  Interventions: Other: Tri-Membrane Wrap™ DFU
- DFU Membrane Wrap™ + SOC (Experimental): Membrane Wrap™ is an allograft derived from human amniotic membrane.
  Interventions: Other: Membrane Wrap™ DFU
- DFU Membrane Wrap-Lite™ + SOC (Experimental): Membrane Wrap-Lite™ is an allograft derived from human amniotic membrane.
  Interventions: Other: Membrane Wrap-Lite™ DFU
- DFU Membrane Wrap-Hydro™ + SOC (Experimental): Membrane Wrap-Hydro™ is an allograft derived from human amniotic membrane.
  Interventions: Other: Membrane Wrap-Hydro™ DFU
- VLU Standard of Care (Active Comparator): Debridement, reduction of bacterial burden, and proper moisture balance using dressings. Compression using multilayer compression wraps.
  Interventions: Other: Standard of Care VLU
- VLU Tri-Membrane Wrap™ + SOC (Experimental): Tri-Membrane Wrap™ is an allograft derived from human amniotic membrane.
  Interventions: Other: Tri-Membrane Wrap™ VLU
- VLU Membrane Wrap™ + SOC (Experimental): Membrane Wrap™ is an allograft derived from human amniotic membrane.
  Interventions: Other: Membrane Wrap™ VLU
- VLU Membrane Wrap-Lite™ + SOC (Experimental): Membrane Wrap-Lite™ is an allograft derived from human amniotic membrane.
  Interventions: Other: Membrane Wrap-Lite™ VLU
- VLU Membrane Wrap-Hydro™ + SOC (Experimental): Membrane Wrap-Hydro™ is an allograft derived from human amniotic membrane.
  Interventions: Other: Membrane Wrap-Hydro™ VLU

INTERVENTIONS:
Other: Standard of Care DFU — Beginning at the screening visit, participants will receive weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: DFU Standard of Care
Other: Tri-Membrane Wrap™ DFU — Participants will receive weekly applications of Tri-Membrane Wrap™ and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: DFU Tri-Membrane Wrap™ + SOC
Other: Membrane Wrap™ DFU — Participants will receive weekly applications of Membrane Wrap™ and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: DFU Membrane Wrap™ + SOC
Other: Membrane Wrap-Lite™ DFU — Participants will receive weekly applications of Membrane Wrap-Lite™ and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: DFU Membrane Wrap-Lite™ + SOC
Other: Membrane Wrap-Hydro™ DFU — Participants will receive weekly applications of Membrane Wrap-Hydro™ and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: DFU Membrane Wrap-Hydro™ + SOC
Other: Standard of Care VLU — Beginning at the screening visit, participants will receive weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and compression) until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: VLU Standard of Care
Other: Tri-Membrane Wrap™ VLU — Participants will receive weekly applications of Tri-Membrane Wrap™ and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: VLU Tri-Membrane Wrap™ + SOC
Other: Membrane Wrap™ VLU — Participants will receive weekly applications of Membrane Wrap™ and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: VLU Membrane Wrap™ + SOC
Other: Membrane Wrap-Lite™ VLU — Participants will receive weekly applications of Membrane Wrap-Lite™ and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: VLU Membrane Wrap-Lite™ + SOC
Other: Membrane Wrap-Hydro™ VLU — Participants will receive weekly applications of Membrane Wrap-Hydro™ and Standard of Care until ulcer closure, or a maximum of 12 weeks, whichever occurs first.
  Arms: VLU Membrane Wrap-Hydro™ + SOC

SUMMARY:
The purpose of this study is to evaluate the efficacy of human placental membrane products and standard of care versus standard of care alone in the management of nonhealing diabetic foot ulcers and venous leg ulcers.

DETAILED DESCRIPTION:
This study is a multi-center, prospective, randomized controlled clinical study consisting of 650 subjects from up to 30 centers. The subjects are randomized to receive 1 of 4 treatments, either with Tri-Membrane Wrap™ (HPM-1); Membrane Wrap™ (HPM-2); Membrane Wrap-Lite™ (HPM-3); Membrane Wrap-Hydro™ (HPM-4); and SOC. The target ulcers are evaluated weekly by the investigator. The subject is treated once a week, to receive weekly applications of HPM-1 - HPM - 4 + SOC or SOC alone until or up to 12 weeks or until the study ulcer has completely closed (i.e. 100% closure as assessed by the investigator and confirmed 2 weeks later at the closure confirmation visit (CCV). One additional visit per week is optional for both arms, for the purpose of changing only (1) the secondary dressing in the HPM arm or (2) change the standard of care dressing in the control arm. A trial design diagram is found in Figure 3.

ELIGIBILITY:
Inclusion Criteria:

* The potential subject must be at least 18 years of age or older.
* The potential subject must have a diagnosis of type 1 or 2 Diabetes mellitus.
* At enrollment, the potential subject must have a target ulcer with a minimum surface area of 1.0 cm2 and a maximum surface area of 20 cm2 measured post debridement with the eKare inSight® imaging device.
* The potential subject must have a target ulcer that has been present for a minimum of 4 weeks of standard of care, prior to the initial screening visit.
* The potential subject must have a target ulcer located on the foot with at least 50% of the ulcer below the malleolus.
* The potential subject must have a target ulcer that is Wagner 1 or 2 grade, extending at least through the dermis or subcutaneous tissue and may involve the muscle provided it is below the medial aspect of the malleolus. The ulcer may not include exposed tendon or bone.
* The potential subject's affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 3 months of the first screening visit are acceptable:

  1. ABI between 0.7 and ≤ 1.3;
  2. TBI ≥ 0.6;
  3. TCOM ≥ 40 mmHg;
  4. PVR: biphasic.
* If the potential subject has two or more ulcers, they must be separated by at least 2 cm. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
* The potential subject must consent to using the prescribed offloading method for the duration of the study.
* The potential subject must agree to attend the weekly study visits required by the protocol.
* The potential subject must be willing and able to participate in the informed consent process.

Exclusion Criteria: DFU

* The potential subject is known to have a life expectancy of < 6 months.
* The potential subject's target ulcer is not secondary to diabetes.
* The target ulcer is infected or there is cellulitis in the surrounding skin.
* The target ulcer exposes tendon or bone.
* There is evidence of osteomyelitis complicating the target ulcer.
* There is an infection in the target ulcer or in a remote location that requires systemic antibiotic therapy.
* The potential subject is receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of prednisone per day or equivalent) or cytotoxic chemotherapy or is taking medications that the PI believes will interfere with wound healing (e.g., biologics).
* The potential subject is taking hydroxyurea.
* The potential subject has applied topical steroids to the ulcer surface within one month of initial screening.
* The potential subject with a previous partial amputation on the affected foot that results in a deformity that impedes proper offloading of the target ulcer.
* The potential subject has glycated hemoglobin (HbA1c) greater than or equal to 12% within 3 months of the initial screening visit.
* The surface area of the potential subject's target ulcer has reduced in size by more than 40% in the 4 weeks prior to Treatment Visit 1 ("historical" run-in period*). OR The surface area of the potential subject's target ulcer has reduced in size by more than 20% in the 2 weeks prior to the initial screening visit AND The surface area measurement of the potential subject's target ulcer decreases by 25% or more during the active 2-week screening phase: the 2 weeks from the initial screening visit (SV1) to the TV-1 visit.

  a. eKare inSight® imaging device is not required for measurements taken during the historical run-in period (e.g., calculating surface area using length X width is acceptable)
* The potential subject has an acute Charcot foot, or an inactive Charcot foot, which impedes proper offloading of the target ulcer.
* The potential subject is a woman who is pregnant or considering becoming pregnant within the next 6 months.
* The potential subject has end stage renal disease requiring dialysis.
* The potential subject has participated in a clinical trial involving treatment with an investigational product within the previous 30 days.
* The potential subject, in the opinion of the investigator, has a medical or psychological condition that may interfere with study assessments.
* The potential subject was treated with hyperbaric oxygen therapy (HBOT) or a Cellular, Acellular, Matrix-like Product (CAMP) in the 30 days prior to the initial screening visit.
* The potential subject has a malnutrition indicator score <17 as measured on the Mini Nutritional Assessment.

Inclusion Criteria:VLU

* The potential subject must be at least 21 years of age or older.
* At enrollment, the potential subjects must have a target ulcer with a minimum surface area of 1 cm2 and a maximum surface area of 20 cm2 measured post-debridement.
* The potential subject must have a target ulcer that has been present for a minimum of 4 weeks of standard of care prior to the initial screening visit.
* The potential subject's affected limb must have adequate perfusion confirmed by vascular assessment. Any of the following methods performed within 3 months of the first screening visit are acceptable:

  1. ABI between 0.7 and ≤ 1.3;
  2. TBI ≥ 0.6;
  3. TCOM ≥ 40 mmHg;
  4. PVR: biphasic.
* If the potential subject has two or more ulcers, they must be separated by at least 2 cm post-debridement. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
* The potential subject must agree to attend the weekly study visits required by the protocol.
* The potential subject must be willing and able to participate in the informed consent process.

Exclusion Criteria:

* The potential subject is known to have a life expectancy of < 6 months.
* The potential subject's target ulcer is infected, requires systemic antibiotic therapy, or there is cellulitis in the surrounding skin.
* The potential subject's target ulcer exposes tendon or bone.
* There is evidence of osteomyelitis complicating the potential subject's target ulcer.
* The potential subject is receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of prednisone per day or equivalent) or cytotoxic chemotherapy or is taking medications that the PI believes will interfere with wound healing (e.g., biologics).
* The potential subject has applied topical steroids to the ulcer surface within one month of initial screening.
* The potential subject has glycated hemoglobin (HbA1c) greater than or equal to 12% within 3 months of the initial screening visit.
* The surface area of the potential subject's target ulcer has reduced in size by more than 40% in the 4 weeks prior to Treatment Visit 1 ("historical" run-in period*). OR The surface area of the potential subject's target ulcer has reduced in size by more than 20% in the 2 weeks prior to the initial screening visit AND The surface area measurement of the potential subject's target ulcer decreases by 25% or more during the active 2-week screening phase: the 2 weeks from the initial screening visit (SV1) to the TV-1 visit.

  a. *eKare inSight® imaging device is not required for measurements taken during the historical run-in period (e.g., calculating surface area using length X width is acceptable)
* The potential subject is a woman who is pregnant or considering becoming pregnant within the next 6 months.
* The potential subject has end stage renal disease requiring dialysis.
* The potential subject has participated in a clinical trial involving treatment with an investigational product within the previous 30 days.
* A potential subject who, in the opinion of the investigator, has a medical or psychological condition that may interfere with study assessments.
* The potential subject was treated with hyperbaric oxygen therapy (HBOT) or a Cellular, Acellular, Matrix-like Product (CAMP) in the 30 days prior to the initial screening visit.
* The potential subject has a malnutrition indicator score <17 as measured on the Mini Nutritional Assessment.
* The potential subject has a wound with active or latent infection.
* The subject has a disorder that would create unacceptable risk of post-operative complication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Determine the between-arm difference percentage of subjects achieving complete closure of target ulcer over 12 weeks. | 1-12 Weeks
  To determine the between-arm difference of multiple Human Placental Membrane (HPM) products plus SOC versus SOC alone in achieving complete closure of nonhealing diabetic foot ulcers and venous leg ulcers over 12 weeks using a modified dual platform (Matriarch) trial design. The initial plan is to evaluate several HPM per wound type; however, the modified platform design permits the inclusion of additional placental and umbilical cord derived products and can continue in perpetuity.

SECONDARY OUTCOMES:
Time to Closure | 1-12 weeks
  To determine the between-arm difference in the time to closure over 12 weeks for HPM plus SOC versus SOC alone.
Percent Area Reduction (PAR) | 1-12 weeks
  To determine the between-arm difference in the percent area reduction (PAR) at weekly intervals for HPM plus SOC versus SOC alone.
Determine improvement in quality of life | 1-12 Weeks
  To determine the between-arm difference in the quality of life for subjects receiving HPM plus SOC compared to SOC alone using the Wound Quality of Life (wQOL) questionnaire. Scores on a scare from "Not at all" to "Very much."
Pain in patients who present with VAS greater than 4 | 1-12 weeks
  To determine the between-arm difference in pain for patients that present with a Visual Analog Sale (VAS) score of greater than 4. The VAS has a scale of 0-10. 0 Meaning no pain and 10 being the worst pain.
Proportion of patients that reach complete closure over 65 | 1-12 weeks
  To determine the proportion of ulcers that heal in patients 65 years or older for HPM plus SOC versus SOC alone.
Functional Ambulatory Category Scale | 1-12 Weeks
  To evaluate the between-arm difference in functional ambulation based on Functional Ambulatory Category Scale (FACS) - VLU subjects only. FACS is a scale from 0-5, 5 being completely independent and ambulatory on all surfaces.
Determine improvement in quality of life | 1-12 Weeks
  To determine the between-arm difference in the quality of life for subjects receiving HPM plus SOC compared to SOC alone using the Forgotten Wound Score (FWS) questionnaire. Forgotten wound scores situations on a scale of "never" to "mostly."

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Foot and Ankle Disorders, Philidelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No